CLINICAL TRIAL: NCT07254897
Title: Long-term Muscle Synthetic Effects of Intradialytic Parenteral Nutrition in Chronic Hemodialysis Patients
Acronym: LOTUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Wesley Visser, Principal investigator, PhD, RD, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-522111-42-02; 2025-522111-42-02 (EU CTIS Number)
Record Dates: First submitted 2025-11-16; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Malnutrition or Risk of Malnutrition
Keywords: hemodialysis; myofibrillar fractional synthetic rate; intradialytic parenteral nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Investigator-initiated intervention study with crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intra dialytic parenteral nutrition (Olimel N12, Baxter, 1L/session) (Experimental): intra dialytic parenteral nutrition (Olimel N12, Baxter, 1L/session)
  Interventions: Dietary Supplement: intra dialytic parenteral nutrition (Olimel N12, Baxter, 1L/session)
- Control (No Intervention): no intervention according to usual care

INTERVENTIONS:
Dietary Supplement: intra dialytic parenteral nutrition (Olimel N12, Baxter, 1L/session) — Olimel N12 is administered via the arteriovenous fistula. Olimel N12 is registered for parenteral use in day-care settings. The dose is 1000 mL (250 mL/h) per hemodialysis session.
  Arms: intra dialytic parenteral nutrition (Olimel N12, Baxter, 1L/session)

SUMMARY:
This study examines the effects of intradialytic parenteral nutrition (IDPN) on muscle growth and blood pressure in patients undergoing chronic hemodialysis.

DETAILED DESCRIPTION:
Rationale: Malnutrition and a negative protein balance are highly prevalent in hemodialysis (HD) patients. In these patients, nutritional status and body composition are closely linked to morbidity, mortality, and quality of life. Muscle wasting in HD patients is the result of poor intake, anabolic resistance and the intradialytic loss of amino acids, leading to a negative protein balance. Intradialytic parenteral nutrition (IDPN) has been shown to reverse this anabolic state in the short term (a single dialysis session) in studies using primed constant infusion of isotope-labeled amino acids. However, such studies were carried out in fasted state, which may significantly overestimate the effect. Moreover, they provide no insight in muscle synthesis over longer periods of time, including the interdialytic interval and across multiple dialysis sessions. The use of deuterated water (2H2O) enables longer-term assessment of muscle protein synthesis in an outpatient setting. The administration of IDPN, due to its volume, may have intradialytic hemodynamic effects, which have not been characterized in previous studies.

Objective: To study the effect of IDPN on muscle protein synthesis in chronic hemodialysis patients and to characterize the hemodynamic effects of IDPN.

Study design: Investigator-initiated intervention study with crossover design.

Study population: Chronic hemodialysis patients aged over 18 years (dialysis vintage over 3 months).

Intervention: IDPN (Olimel N12, Baxter, 1L/session) or regular care without IDPN.

Main study parameters/endpoints: Difference in myofibrillar fractional synthetic rate during a one-week treatment with IDPN versus one control week consisting of regular care.

Data collection: The study includes a maximum of 9 study visits, which will take place during regular hemodialysis sessions. These may include non-invasive measurements such as bioimpedance spectroscopy, measurements of cardiac output, blood sampling (for which venepuncture), three percutaneous muscle biopsies (vastus lateralis), food intake registration, collection of dialysate, handgrip strength and activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Receiving HD treatment over 3 months
* Receiving HD treatment 3 times per week for at least 4 hours per session
* 24-hour urine production < 100 mL
* Adequate dialysis dose (eKt/V over 1.2)
* AV fistula with blood flow (measured invasively or by Doppler ultrasound) over 750 mL/min

Exclusion Criteria:

* Occurrence of intradialytic hypotension in the last month, defined by systolic blood pressure < 90 mm Hg combined with a nursing intervention
* Hospitalization < 3 months before inclusion
* Active infection or inflammation at randomization
* Use of oral or intravenous corticosteroids
* Incapacitation
* Patients who are not expected to be able to complete the study protocol (e.g., due to a planned kidney transplantation within the planned study time frame)
* Pregnancy
* Use of oral anticoagulants or antiplatelet agents that cannot be safely stopped during the study
* Diabetes mellitus
* AV fistula with recirculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar fractional synthetic rate | At baseline and during the first dialysis sessions in the following two weeks.
  Difference in myofibrillar fractional synthetic rate during treatment with IDPN versus usual care

SECONDARY OUTCOMES:
Forearm amino acid (AA) balance | During the first visit in intervention and cross-over usual care regiment.
  A cannula is placed in the antecubital vein of the arm opposite the hemodialysis AV fistula. Blood is drawn before hemodialysis, after 2 hours, and at the end of the session from both the cannula (draining forearm musculature) and the "arterial" needle in the AV fistula (representing arterial blood). The "venous" needle is used for infusion. Blood flow and recirculation are checked to prevent mixing of IDPN/placebo-infused blood. Comparing amino acid concentrations before and after the forearm musculature reveals the net uptake or release from the arm.
Intradialytic blood pressure and cardiac output | Cardiac output will be measured at baseline and during the first dialysis sesions in the following 2 weeks. Predialysis systolic blood pressure, intradialytic blood pressure decrease, and ultrafiltration volume will be measured at each dialysis session.
  Cardiac output can be estimated noninvasively by the Starling Monitor (Baxter). This method relies on bioreactance measured by 4 electrodes placed on the patient's chest. By employing this method, cardiac output can be measured continuously with no disruption to the treatment and no discomfort to the patient. Predialysis systolic blood pressure, intradialytic blood pressure decrease, and ultrafiltration volume will be assessed.
Amino acid loss in dialysate | Amino acid loss in dialysate will be measured during V2 and V5.
  During hemodialysis, some AA are lost in the dialysate. This amount is likely to increase during IDPN, given the significantly elevated plasma AA concentrations during this treatment. To quantify this, we will collect all spent dialysate in a specially constructed collection device.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No